CLINICAL TRIAL: NCT00382967
Title: A Multicentre, Randomised, Open Label, Comparative Phase 4 Trial to Assess Changes in Clinical Management After DaTSCAN Imaging of Subjects With Clinically Uncertain Parkinsonism in a General Neurologist Setting.
Brief Title: A Study to Assess Changes in Clinical Management After DaTSCAN Imaging of Subjects With Clinically Uncertain Parkinsonism or an Illness With Similar Symptoms
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GE Healthcare (Industry)
Collaborators: i3 Statprobe (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDT409
Record Dates: First submitted 2006-09-29; First posted 2006-10-02 (Estimated); Results first posted 2012-08-29 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Parkinsonian Syndromes
Keywords: Parkinsonian Syndromes, Parkinsonism, DaTSCAN, SPECT, clinical management, quality of life, movement disorder; Clinically uncertain Parkinsonian Syndromes
MeSH Terms: conditions — Parkinsonian Disorders; Movement Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Datscan Product (Experimental)
  Interventions: Procedure: DaTSCAN SPECT imaging
- Control (No Intervention)

INTERVENTIONS:
Procedure: DaTSCAN SPECT imaging — A single intravenous injection of DaTSCAN with a total activity of 111-185 MBq (volume of 2.5 or 5.0 mL). SPECT scanning to be performed 3 to 6 hours after DaTSCAN injection.
  Other Names: I-123 Ioflupane
  Arms: Datscan Product

SUMMARY:
Patients come to their doctor showing possible symptoms of a movement disorder. It is possible that these symptoms may get worse over time. There is more than one disease that can cause such symptoms. The most common movement disorder illnesses are Parkinson´s Disease and Essential Tremor. Sometimes it is difficult for doctors to make the right diagnosis because the symptoms caused by these illnesses are almost the same. On the other hand the correct treatment for Parkinson´s Disease is different from the correct treatment for Essential Tremor. This study aims to see whether having pictures of the brain taken with DaTSCAN can affect the way the doctor treats these patients and whether it can affect their quality of life directly.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with clinically uncertain Parkinsonian Syndromes or monosymptomatic, atypical or incomplete presentation of tremor, rigidity, bradykinesia or postural instability.
* Onset of clinical manifestations within the last 5 years

Exclusion Criteria:

* Differential diagnosis between Parkinsons´s Disease and Progressive Supranuclear Palsy or between Parkinson´s Disease and Multiple System Atrophy
* Subjects with an established/certain movement disorder clinical diagnosis
* Presence of known causes of tremor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 273 (Actual)
Dates: Start 2006-10; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Andreas Kupsch, Principal Investigator — Virchov Klinikum, Berlin, Germany; Paul Sherwin, MD, Study Director — GE Healthcare
Locations (2):
- GE Healthcare, Princeton, New Jersey, United States
- GE Healthcare, Vélizy-Villacoublay, France

REFERENCES:
- [Derived] Kupsch AR, Bajaj N, Weiland F, Tartaglione A, Klutmann S, Buitendyk M, Sherwin P, Tate A, Grachev ID. Impact of DaTscan SPECT imaging on clinical management, diagnosis, confidence of diagnosis, quality of life, health resource use and safety in patients with clinically uncertain parkinsonian syndromes: a prospective 1-year follow-up of an open-label controlled study. J Neurol Neurosurg Psychiatry. 2012 Jun;83(6):620-8. doi: 10.1136/jnnp-2011-301695. Epub 2012 Apr 6. PMID 22492213

RESULTS

PARTICIPANT FLOW:
Groups:
- Datscan Product: [Iodine-123]Ioflupane isotonic solution. Single i.v. injection within the dose range of 111 to 185 Megabecquerel (MBq) [3-5 millicurie (mCi)].
- Control Arm: No (Injection) Intervention
Period: Overall Study
Arm/Group | Datscan Product | Control Arm
Started | 122 (135 subjects enrolled at the start of the study, however, 13 subjects withdrew prior to dosing.) | 138
Completed | 121 (Patient lost to followup and the data was not recorded.) | 137 (Subject dosed in error, should not have received Datscan product)
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Datscan Product | Control Arm | Total
Number analyzed (Participants) | 121 | 137 | 258
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 55 | 101
  >=65 years | 75 | 82 | 157
Age Continuous [Mean (Standard Deviation); unit: years] | 66.9 (12.1) | 65.5 (11.8) | 66.2 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 63 | 119
  Male | 65 | 74 | 139
Region of Enrollment [Number; unit: participants]
  United States | 32 | 37 | 69
  France | 2 | 2 | 4
  Denmark | 2 | 2 | 4
  Germany | 20 | 20 | 40
  Italy | 12 | 14 | 26
  Norway | 8 | 8 | 16
  Spain | 6 | 11 | 17
  Switzerland | 1 | 2 | 3
  United Kingdom | 38 | 41 | 79

OUTCOME MEASURES:

1. Primary Outcome: Changes That the Doctor Made in the Clinical Management of Subjects Based Upon the Impact of the Imaging Product.
Description: The impact the Datscan image had on the Doctor's decisions on the clinical management of subjects. A record of the number of changes in the Doctor's clinical management. It is possible for a subject to have multiple changes in Clinical management and other subjects to have no change in their management.
Time Frame: Changes in clinical management made from Visit 1 (baseline) to Visit 3 (a 3 month period)
Measure: Number; unit: Number of changes in clinical management
Arm/Group | Datscan Product | Control Arm
Number analyzed (Participants) | 116 | 128
Number of changes in clinical management
  Initiation of medication not planned | 33 | 28
  Avoidance/withdrawal of medication planned | 19 | 11
  Performance of diagnostic test not planned | 6 | 6
  Avoidance of diagnostic test planned | 1 | 0
  Arrangement of a referral not planned | 4 | 2
  Cancellation of a referral planned | 0 | 0
  Other Actions | 16 | 6
  Significant changes made | 58 | 40

2. Secondary Outcome: Changes That the Doctor Made in the Clinical Management of Subjects Based Upon the Impact of the Imaging Product.
Description: The impact the Datscan image had on the Doctor's decisions on the clinical management of subjects. A record of the number of changes in the Doctor's clinical management. From the first patient visit (baseline) to the fourth patient visit, which was 12 months. This was a 1 year time period being assessed.It is possible for a subject to have multiple changes in Clinical management and other subjects to have no change in their management.
Time Frame: From the first patient Visit 1 (1 month) to Visit 4 (12 months). This goes from the baseline (visit 1) up to 1 year post contrast administration.
Population: The numbers represent the number of changes in decisions that the Doctor made in the clinical management of the patient with Clinically Uncertain Parkinsonism
Measure: Number; unit: Number of changes in clinical management
Arm/Group | Datscan Product | Control Arm
Number analyzed (Participants) | 116 | 128
Number of changes in clinical management
  Initiation of Medication not planned | 35 | 22
  Avoidance or withdrawal of medication planned | 16 | 6
  Performance of diagnostic test not planned | 7 | 5
  Avoidance of diagnostic test planned | 0 | 0
  Arrangement of referral not planned | 3 | 1
  Cancellation of referral planned | 0 | 1
  Other Actions | 15 | 9
  Significant changes made | 48 | 28

ADVERSE EVENTS:
Arm/Group | Datscan Product | Control Arm
Serious Adverse Events (participants affected / at risk) | 0/122 | 0/137
Other Adverse Events (participants affected / at risk) | 0/122 | 0/137

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No